CLINICAL TRIAL: NCT07104006
Title: Development and Testing of a Smoking Cessation Intervention Using Multi-Theory Model (MTM) Among Young Adults: A Randomized Controlled Trial
Brief Title: Smoking Cessation Intervention for Young Adults Using MTM: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Timothy Grigsby, Assistant Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB #: UNLV-2025-174
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Tobacco Use Disorder/Cigarette Smoking
Keywords: Smoking cessation intervention; Multi-Theory Model (MTM) of Behavior Change; Young adults; Randomized controlled trial (RCT)
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking; Myopathies, Structural, Congenital

STUDY DESIGN:
Intervention Model Description: This study is a two-arm randomized controlled trial (RCT) designed to evaluate the effectiveness of a smoking cessation intervention based on the Multi-Theory Model (MTM) among young adults aged 18-29. Participants are randomly assigned to either the MTM-based intervention group or a control group receiving knowledge based intervention. The intervention is delivered exclusively online to optimize accessibility, participant engagement, and scalability. The MTM framework guides behavior change strategies focused on both initiation and maintenance of smoking cessation. Outcomes are measured at baseline, immediately post-intervention, and at 12-week follow-up to assess efficacy and sustainability of quitting behaviors. Individual-level randomization minimizes contamination between groups and strengthens internal validity by ensuring balanced allocation of participants across intervention and control arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knowledge-Based Smoking Risk Education and Quit Strategies (Active Comparator): Participants are individually randomized to the control arm receive a four-week educational program focusing on basic information about the health risks of smoking and effective quitting techniques. The program consists of weekly 90-minute sessions delivered in an online format to maximize participant reach and accessibility. Sessions cover topics such as smoking-related health consequences, benefits of quitting, common barriers to cessation, and practical strategies for quitting smoking. Unlike the experimental arm, this program does not include behavior change techniques grounded in the Multi-Theory Model but instead emphasizes increasing awareness and knowledge to motivate cessation. This active comparator arm serves to control for time and attention while providing participants with standard smoking cessation information.
  Interventions: Behavioral: Multi-Theory Model (MTM)-Based Smoking Cessation Program
- Multi-Theory Model-Based Smoking Cessation Intervention (Experimental): This arm delivers a four-week smoking cessation intervention grounded in the Multi-Theory Model (MTM) of health behavior change. Participants are individually randomized into two arms of the study to ensure comparability between groups and reduce selection bias. The intervention comprises weekly 90-minute sessions delivered entirely online, with a focus on core MTM constructs: participatory dialogue, behavioral confidence, emotional transformation, practice for change, and changes in physical and social environment.
  Session activities include storytelling, interactive discussions weighing quitting pros and cons, confidence-building exercises, role-playing high-risk situations, emotional expression and transformation techniques, development of supportive social networks, stress management tools, reflection and reward practices, and commitment reinforcement through letters and group sharing.
  Interventions: Behavioral: Multi-Theory Model (MTM)-Based Smoking Cessation Program

INTERVENTIONS:
Behavioral: Multi-Theory Model (MTM)-Based Smoking Cessation Program — Multi-Theory Model (MTM)-Based Smoking Cessation Program: A four-week online smoking cessation program based on the Multi-Theory Model (MTM). It uses behavior change strategies including participatory dialogue, building confidence, emotional transformation, practice for change, and changes in physical and social environment. Activities include storytelling, role-playing high-risk situations, emotional regulation, social support, stress management, reflection, and commitment exercises. The goal is to help young adults initiate and maintain quitting smoking.
  Knowledge-Based Smoking Risk Education and Quit Strategies Program: A four-week, online educational program providing information on smoking risks, benefits of quitting, barriers, and practical quit strategies. This control arm focuses on increasing knowledge and awareness but does not include MTM-based behavior change techniques.

SUMMARY:
The goal of this clinical trial is to evaluate whether a Multi-Theory Model (MTM)-based behavioral intervention can effectively promote smoking cessation and support behavior change in young adult cigarette smokers aged 18 to 29 in the United States. This trial focuses on whether applying theory-driven strategies such as emotional transformation, behavioral confidence, and participatory dialogue can lead to higher smoking abstinence rates and improved psychosocial outcomes compared to a standard knowledge-based smoking education control group.

The main questions it aims to answer are:

* Does the intervention lead to a greater reduction in nicotine dependence scores (measured by the Fagerström Test for Nicotine Dependence [FTND]) and an increase in quit rate among young adult smokers from baseline to 12-week follow-up?
* Does the MTM-based intervention significantly improve 7-day point prevalence abstinence (PPA) at 12 weeks compared to a knowledge-based control group?
* Does the intervention result in significant positive changes in MTM constructs such as participatory dialogue, behavioral confidence, emotional transformation, practice for change, and changes in the physical and social environment from baseline to 12-week follow-up? Researchers will compare the MTM-based intervention group (experimental arm) to a knowledge-based smoking education control group to determine whether the theory-driven program is more effective in supporting smoking cessation and behavior change among young adult smokers.

Participants will:

* Complete surveys at three time points: baseline (Week 0), post-intervention (Week 5), and follow-up (Week 12), covering demographics, smoking history, nicotine dependence (FTND), MTM constructs (via a validated 48-item scale), and self-reported quit rates.
* Be randomly assigned to one of two groups:

  o MTM-Based Intervention Group: Attend four weekly 90-minute virtual group sessions covering: Week 1: Participatory dialogue, behavioral confidence, and process evaluation Week 2: Emotional transformation, environmental restructuring, and process evaluation Week 3: Practice for change, relapse prevention, and process evaluation Week 4: Social support, reward systems, and process evaluation

  o Knowledge-Based Control Group: Attend four weekly 90-minute didactic virtual sessions focused on: Smoking-related health risks Overview of FDA-approved smoking cessation tools
* Undergo process evaluations using the RQFSM model (Reach, Quality, Fidelity, Satisfaction, and Management) at the end of the intervention to assess how well each program was delivered and perceived.
* Have the optional opportunity for biochemical verification of smoking abstinence using exhaled carbon monoxide (CO) testing.

This trial will be conducted entirely online and follows a randomized controlled trial (RCT) design with a 1:1 group allocation ratio. A total of 144 participants (approximately 72 per group) will be recruited, accounting for an expected attrition rate of up to 50%. This sample size was chosen to ensure sufficient power to detect statistically significant differences between the two groups (effect size f = 0.25, α = 0.05, power = 0.80).

Although the intervention will be delivered virtually, the study is affiliated with the University of Nevada, Las Vegas (UNLV), which provides IRB approval, secure data storage infrastructure, and institutional oversight (IRB Protocol #2024-453). Informed consent will be obtained electronically, and all participant data will be securely stored using encrypted Qualtrics surveys and password-protected UNLV or Google Drive servers with limited access, ensuring full confidentiality and ethical compliance.

This trial addresses a pressing public health challenge: the persistent difficulty young adults face in quitting smoking despite decades of tobacco control efforts. Young adults remain a high-risk population for relapse and are frequently underserved by conventional cessation programs. This MTM-based intervention seeks to fill this gap by targeting both behavioral and environmental barriers through structured, evidence-based strategies designed to build self-efficacy, emotional readiness, and environmental support.

The use of MTM constructs such as emotional transformation, behavioral confidence, and restructuring the physical/social environment is a key innovation that may enhance long-term cessation outcomes. Moreover, delivering the program virtually increases its potential for scalability and real-world application, making it a promising model for public health programs nationwide.

The findings of this clinical trial will be disseminated through peer-reviewed journal articles, national public health conferences (APHA, SOPHE etc.), and shared with stakeholders like the CDC's Office on Smoking and Health. The results may help shape future funding priorities, guide the development of policy, and inform the design of tailored interventions for smoking cessation among young adults.

DETAILED DESCRIPTION:
1. Introduction Tobacco use continues to be a major contributor to preventable disease, disability, and death worldwide. In the United States, despite a general decline in smoking prevalence over the past decades, young adults aged 18-29 continue to demonstrate concerning rates of smoking initiation and persistent use. According to the CDC (2022), approximately 13.8% of individuals in this age group are current cigarette smokers. This prevalence underscores the urgent need for tailored, developmentally appropriate interventions.

   Young adulthood is a transitional period marked by increased autonomy, identity exploration, and greater susceptibility to risk-taking behaviors. These developmental vulnerabilities are compounded by stress, peer influence, and underdeveloped coping mechanisms, making smoking both an appealing coping strategy and a challenging habit to break. Many young adults begin smoking due to social pressures or emotional distress and struggle to quit due to nicotine addiction, insufficient resources, or low behavioral confidence. Alarmingly, although 67.7% of young adult smokers express a desire to quit, only 8.8% successfully do so.

   Smoking-related illnesses claim more than 480,000 lives annually in the U.S. and afflict over 16 million people. Globally, over 1.3 billion people use tobacco, with young adults comprising a substantial proportion. In the U.S., daily smoking among young adults rose from 38.7% to 55.9%, and initiation rates climbed from 20.6% in 2002 to 42.6% in 2018. Disparities are even more severe among marginalized groups including low-income populations, racial/ethnic minorities, and LGBTQ+ individuals due to factors like targeted tobacco marketing, limited access to culturally sensitive care, and socioeconomic barriers.

   Multiple factors contribute to sustained tobacco use among young adults. Biologically, neurodevelopmental immaturity and genetic predisposition increase susceptibility to nicotine addiction. Psychologically, factors such as anxiety, depression, impulsivity, and stress drive smoking behavior. Social influences including peer norms and social modeling strongly affect initiation and continuation. Environmental exposures to tobacco advertising and inadequate policy enforcement further exacerbate these risks.

   The short- and long-term health consequences of smoking are well-documented. Acute effects include impaired lung function, increased heart rate, and elevated blood pressure. Chronic exposure leads to diseases such as COPD, cardiovascular disease, and various cancers. Reproductive health is also compromised, with links to infertility and pregnancy complications.

   Moreover, smoking exacerbates mental health conditions and impairs stress coping. Despite the known risks, many young adults lack access to evidence-based, culturally relevant, and behaviorally grounded cessation interventions. Existing programs often rely on outdated models developed for adolescents or older adults, failing to meet the psychological and contextual needs of younger populations. Although digital platforms offer new opportunities, high attrition rates and lack of theoretical grounding limit their effectiveness.
2. Background and Rationale

   2.1 Public Health Significance Tobacco-related illness remains a leading cause of preventable death in the U.S., with substantial social and economic burdens. Intervening in young adulthood, before lifelong patterns are firmly established, presents a crucial opportunity to reduce future morbidity and mortality.

   2.2 Theoretical Framework While traditional behavioral models like the Transtheoretical Model (TTM), Social Cognitive Theory (SCT), and Health Belief Model (HBM) have been widely used in cessation programs, they often treat behavior change as linear or static. These limitations reduce their effectiveness in addressing the fluctuating motivations and emotional stressors common among young adults.

   This study utilizes the Multi-Theory Model (MTM) of Health Behavior Change, a dynamic and integrative framework that distinguishes between initiation and sustenance phases. MTM constructs include participatory dialogue (weighing pros and cons), behavioral confidence (akin to self-efficacy), changes in the physical environment, emotional transformation, practice for change, and restructuring the social environment. MTM has demonstrated effectiveness in various public health contexts and is particularly well-suited to the diverse and evolving behavioral patterns of young adults.

   2.3 Evidence Gap Despite MTM's theoretical promise, its application to smoking cessation in young adults is limited. Most available programs fail to incorporate emotional regulation, peer support, or environmental restructuring components that are central to sustained behavior change in this age group. Furthermore, culturally and developmentally tailored interventions remain scarce, leaving many at-risk young adults underserved. This study represents one of the first attempts to systematically apply and evaluate MTM constructs in a targeted smoking cessation intervention for this population.

   By designing an MTM-based intervention specifically for young adults, this research aims to fill a critical gap in the public health literature and contribute a replicable, theory-driven model for future cessation programs.
3. Study Objectives

   3.1 Primary Objectives
   * To determine whether the MTM-based intervention significantly improves 7-day point prevalence abstinence (PPA) at the 12-week follow-up compared to a knowledge-based control group among young adult cigarette smokers.
   * To assess whether the MTM-based intervention leads to a greater reduction in nicotine dependence, as measured by the Fagerström Test for Nicotine Dependence (FTND), compared to the control group.

   3.2 Secondary Objectives
   * To examine the extent to which the intervention results in significant positive changes in Multi-Theory Model (MTM) constructs, including participatory dialogue, behavioral confidence, emotional transformation, practice for change, and modifications in the physical and social environment, from baseline to 12-week follow-up.
   * To assess whether the MTM-based intervention leads to an increase in smoking quit rates among young adult smokers from baseline to the 12-week follow-up.
4. Study Design This study utilizes a two-arm, parallel-group randomized controlled trial (RCT) design to rigorously assess the effectiveness of a Multi-Theory Model (MTM)-based behavioral intervention compared to a knowledge-based smoking cessation intervention. The trial will be entirely conducted online through secure digital platforms (Qualtrics). This fully virtual format was chosen to enhance participant accessibility, especially for geographically diverse populations, and to optimize participant retention over the study duration. The RCT design adheres to CONSORT guidelines for non-pharmacological trials, providing a robust methodological framework for evaluating behavioral interventions.

   Eligible participants will be randomized at the individual level in a 1:1 ratio to one of two intervention arms: (1) an MTM-based behavioral intervention (experimental group) or (2) a knowledge-based control intervention. Randomization will be implemented using a computer-generated allocation sequence with block sizes of four, ensuring balanced group assignment. Stratification by gender and baseline nicotine dependence will be considered to control for potential confounding.

   The intervention period spans four consecutive weeks, during which participants will attend one 90-minute session per week. All sessions will be delivered via encrypted Google Meet to ensure confidentiality and standardization across groups.
5. Intervention Arms

   5.1 MTM-Based Intervention (Experimental Group) The experimental condition is informed by the Multi-Theory Model of Health Behavior Change (MTM), which includes both initiation and sustenance constructs. The intervention content was developed in alignment with validated MTM constructs, incorporating participatory pedagogy and cognitive-behavioral strategies. Each weekly session will be co-facilitated by a trained public health graduate student under supervision of academic advisor. A process evaluation will be conducted at the end of each session using the Reach, Quality control, Fidelity, Satisfaction and Management (RQFSM).

   Session Overview:
   * Week 1: Focus on participatory dialogue and behavioral confidence. Activities include small group discussions, personal reflection worksheets, and confidence-building role-play exercises + process evaluation
   * Week 2: Emphasis on emotional transformation and restructuring physical environments. Participants will learn emotional regulation techniques such as guided imagery and design personalized smoke-free action plans + process evaluation
   * Week 3: Practice for change and relapse prevention strategies. This includes identifying triggers, coping mechanisms, and setting SMART goals + process evaluation
   * Week 4: Social support and reinforcement systems. Group exercises will include buddy systems, social media support groups, and reward tracking + process evaluation

   5.2 Knowledge-Based Intervention (Control Group) Participants in the control group will receive didactic information on smoking cessation strategies, mimicking standard public health education. Content is aligned with U.S. Public Health Service guidelines on tobacco treatment but excludes MTM-based constructs.

   Session Overview:
   * Week 1: Education on the health risks of cigarette smoking, including short-term and long-term consequences.
   * Week 2: Overview of FDA-approved cessation tools, including nicotine replacement therapy (NRT), bupropion, and varenicline.
   * Week 3: Behavioral tips for quitting, including setting a quit date, avoiding triggers, and managing withdrawal symptoms.
   * Week 4: Maintenance strategies and referral to additional cessation resources, including 1-800-QUIT-NOW and Smokefree.gov.
6. Sample Size Calculation Using G*Power 3.1.9.7, a sample size of 144 participants (72 per group) was determined to achieve 80% power to detect a medium effect size (f = 0.25) at a significance level of 0.05 for repeated measures. The calculation accounts for an estimated attrition rate of up to 50%, consistent with online behavioral intervention studies targeting young adults.
7. Randomization and Blinding Randomization will be conducted at the individual level using a computer-generated algorithm with block sizes of four to ensure balanced allocation across study arms. Due to the inherent nature of behavioral interventions, blinding of participants, outcome assessors, and statisticians will not be feasible; however, rigorous standardized protocols will mitigate potential bias in outcome assessment and data analysis.
8. Compensation: Each participant will receive a $10 Amazon e-gift card after completing each of the four intervention sessions, with an additional $10 awarded upon completing the 12-week follow-up assessment, for a total of up to $50. Participants who do not complete all sessions will receive partial incentives based on their level of participation. These incentives are not funded by any external organization or grant but are personally covered by the co-investigator as part of fulfilling the requirements for his doctoral degree.

   Amazon e-gift cards were selected as incentives because they offer a convenient, digital delivery method that aligns with our online intervention. Importantly, Amazon does not sell tobacco products, which helps promote a smoke-free lifestyle and reinforces participants' commitment to quitting. This choice also minimizes logistical barriers while supporting the study's health objectives.
9. Data Collection and Management

   9.1 Timepoints:
   * T0 (Baseline): Demographics, smoking history, MTM construct scores, FTND
   * T1 (Post-Intervention): MTM construct scores, FTND, 7-day PPA, quit rate
   * T2 (12-Week Follow-Up): FTND, 7-day PPA, quit rate, MTM scores

   9.2 Data Collection Tools: All instruments will be administered through Qualtrics, a Health Insurance Portability and Accountability Act (HIPAA)-compliant survey platform. Instruments include (49 items in total):
   * MTM 28-item scale (validated with Cronbach's α > 0.80)
   * FTND (6-item instrument, score range: 0-10)
   * Single-item self-efficacy scale for quit rate: "How confident are you that you can remain completely smoke-free for the next 30 days?" (1 = Not at all confident to 5 = Extremely confident)

   9.3 Data Management: Data will be stored on UNLV's secure, encrypted servers and accessed only by authorized research personnel. Each participant will be assigned a unique identifier to ensure anonymity. Weekly data integrity checks and compliance with General Data Protection Regulation (GDPR) and HIPAA standards will be ensured.

   9.4 Missing Data: Missing data will be handled using Multiple Imputation (MI) under the assumption of Missing at Random (MAR).
10. Ethical Considerations The study protocol has submitted for the approval from the University of Nevada, Las Vegas Institutional Review Board (IRB Protocol #2024-453). Electronic informed consent will be obtained from all participants prior to enrollment. Participants will be informed of their right to withdraw at any time without penalty. All procedures will comply with the Declaration of Helsinki and federal regulations on human subject's research.
11. Dissemination Plan

    Research findings will be shared with both academic and public health audiences. Planned dissemination channels include:
    * Peer-reviewed publications in journals such as Tobacco Control, Nicotine & Tobacco Research, and American Journal of Public Health
    * Conference presentations (e.g., American Public Health Association [APHA], Society for Public Health Education [SOPHE])
    * Policy briefs and executive summaries provided to the Centers for Disease Control and Prevention (CDC) and state/local health departments
    * Lay summaries disseminated via social media platforms and institutional press releases to enhance public engagement
12. Expected Impact This study will contribute new empirical evidence on the utility of the Multi-Theory Model as a framework for behavior change among young adult smokers. By leveraging a fully online design, the intervention could be adapted for national scale-up, particularly among underserved populations with limited access to in-person cessation programs. Findings are expected to inform clinical guidelines, public health curricula, and tobacco control policies aimed at reducing smoking prevalence in young adult populations.

Moreover, the integration of behavior change theory with digital health interventions aligns with national strategic priorities in tobacco control, such as those outlined in the FDA's Comprehensive Plan for Tobacco and Nicotine Regulation and the Healthy People 2030 objectives.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-29 years
* Current smoker (defined as having smoked at least one cigarette daily over the past 7 days)
* Resident of the United States
* Able to read and understand English

Exclusion Criteria:

* Use of non-cigarette tobacco products (e.g., vaping, smokeless tobacco)
* Participation in any other smoking cessation program
* Pregnant or planning to become pregnant during the study period
* Dual or poly-substance users, including alcohol or illicit drugs.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Fagerström Test for Nicotine Dependence (FTND) measure | Baseline to 12 week followup
  This outcome measures changes in nicotine dependence using the Fagerström Test for Nicotine Dependence (FTND), a validated 6-item questionnaire assessing the intensity of physical addiction to nicotine. Scores range from 0 to 10, with higher scores indicating greater dependence. Participants complete the FTND at baseline (pre-intervention) and again at the 12-week follow-up. The difference in scores over time is used to evaluate whether the intervention reduces nicotine dependence among young adult smokers. This helps assess the impact of the intervention beyond smoking cessation, providing insight into reductions in the psychological and physiological aspects of tobacco addiction.
  Repeated Measures Analysis of Covariance (ANCOVA) will be used to examine changes in continuous outcomes (e.g., MTM construct scores, FTND scores) across the three time points. Baseline values and individual-level covariates (e.g., age, gender, baseline dependence) will be included as covariates.
7-day point prevalence abstinence (PPA) | 12-week follow-up after baseline assessment
  The 7-day point prevalence abstinence (PPA) measures whether participants have refrained from smoking defined as no tobacco use, not even a single puff during the 7 days prior to the 12-week follow-up. This outcome is assessed through participant self-report using a standardized questionnaire. To enhance accuracy, abstinence may be optionally validated using a carbon monoxide (CO) breath analyzer, with CO levels ≤6 parts per million (ppm) indicating non-smoking status. This measure helps determine the short-term effectiveness of the intervention in promoting smoking cessation among young adults.

SECONDARY OUTCOMES:
Changes in mean scores of MTM constructs using a validated 28-item MTM instrument | Time of enrollment to 12 week followup
  This outcome measures changes in participants' behavioral and psychological readiness to quit smoking using a validated 28-item questionnaire based on the Multi-Theory Model (MTM) of health behavior change. The instrument assesses six key MTM constructs: participatory dialogue, behavioral confidence, changes in the physical environment, emotional transformation, practice for change, and changes in the social environment. Each construct is measured using a set of Likert-scale items (e.g., 1 = Not at all sure to 5 = Completely sure). Participants complete the survey at baseline, immediately after the 4-week intervention, and at a 12-week follow-up. Mean scores are calculated for each construct at each time point to assess changes in smoking-related beliefs and behaviors over time.
  Generalized Linear Mixed Models (GLMM) with a logit link will assess differences in binary outcomes (PPA and quit rates) over time, incorporating fixed effects for group, time, and group × time interaction.
Quit rate | Baseline to 12-week follow-up
  This outcome measures the self-reported quit rate, defined as the proportion of participants who successfully refrained from smoking for at least 24 consecutive hours with the intention of permanent cessation. Participants are asked whether they made any such quit attempts during the entire study period, particularly between baseline and the 12-week follow-up. A quit attempt is considered valid only if it reflects a deliberate and conscious effort to quit smoking entirely. This measure provides meaningful insight into participants' motivation and readiness to quit, even if sustained abstinence was not achieved. Tracking 24-hour quit rates at follow-up enables evaluation of the behavioral impact of the intervention on smoking cessation efforts among young adults.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nevada, Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified and aggregate-level data will be shared, including summary statistics such as group mean changes, average age, and proportions by gender and other relevant characteristics. This may include aggregated MTM construct scores, smoking status, quit attempts, and 7-day point prevalence abstinence outcomes. Data will be shared for academic research and secondary analysis to promote transparency and advance understanding of smoking cessation interventions. All personal identifiers will be removed to protect confidentiality. IPD will be made available upon reasonable request following publication of the primary results and with approval from the principal investigator and institutional review board (IRB).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: June 2026, for 3 years
Access Criteria: Qualified researchers affiliated with academic institutions or public health organizations may request access to these de-identified, aggregate-level data and supporting materials such as study protocols, data dictionaries, and analysis plans. Access will be granted for non-commercial, scholarly research following submission of a formal proposal outlining study aims and analysis plans. Approval from the principal investigator and the institutional review board (IRB) may be required.
  Upon approval, data will be shared via a secure platform or encrypted file transfer to maintain confidentiality and data integrity. All recipients must sign a data use agreement prohibiting any attempt to re-identify participants or redistribute the data.

REFERENCES:
- [Background] Zhou X, Wei X, Cheng A, Liu Z, Su Z, Li J, Qin R, Zhao L, Xie Y, Huang Z, Xia X, Liu Y, Song Q, Xiao D, Wang C. Mobile Phone-Based Interventions for Smoking Cessation Among Young People: Systematic Review and Meta-Analysis. JMIR Mhealth Uhealth. 2023 Sep 12;11:e48253. doi: 10.2196/48253. PMID 37706482
- [Background] Schnoll RA, Johnson TA, Lerman C. Genetics and smoking behavior. Curr Psychiatry Rep. 2007 Oct;9(5):349-57. doi: 10.1007/s11920-007-0045-3. PMID 17915073
- [Background] Rigotti NA, DiFranza JR, Chang Y, Tisdale T, Kemp B, Singer DE. The effect of enforcing tobacco-sales laws on adolescents' access to tobacco and smoking behavior. N Engl J Med. 1997 Oct 9;337(15):1044-51. doi: 10.1056/NEJM199710093371505. PMID 9321533
- [Background] Ravi K, Indrapriyadharshini K, Madankumar PD. Application of Health Behavioral Models in Smoking Cessation - A Systematic Review. Indian J Public Health. 2021 Apr-Jun;65(2):103-109. doi: 10.4103/ijph.IJPH_1351_20. PMID 34135176
- [Background] Liu ST, Snyder K, Tynan MA, Wang TW. Youth Access to Tobacco Products in the United States, 2016-2018. Tob Regul Sci. 2019 Nov;5(6):491-501. doi: 10.18001/TRS.5.6.2. PMID 31745494
- [Background] Green R, Meredith LR, Mewton L, Squeglia LM. Adolescent Neurodevelopment Within the Context of Impulsivity and Substance Use. Curr Addict Rep. 2023 Jun;10(2):166-177. doi: 10.1007/s40429-023-00485-4. Epub 2023 May 2. PMID 38009082
- [Background] Chen-Sankey JC, Unger JB, Bansal-Travers M, Niederdeppe J, Bernat E, Choi K. E-cigarette Marketing Exposure and Subsequent Experimentation Among Youth and Young Adults. Pediatrics. 2019 Nov;144(5):e20191119. doi: 10.1542/peds.2019-1119. PMID 31659003
- [Background] Chassin L, Presson CC, Pitts SC, Sherman SJ. The natural history of cigarette smoking from adolescence to adulthood in a midwestern community sample: multiple trajectories and their psychosocial correlates. Health Psychol. 2000 May;19(3):223-31. PMID 10868766
- [Background] Brown RA, Abrantes AM, Minami H, Prince MA, Bloom EL, Apodaca TR, Strong DR, Picotte DM, Monti PM, MacPherson L, Matsko SV, Hunt JI. Motivational Interviewing to Reduce Substance Use in Adolescents with Psychiatric Comorbidity. J Subst Abuse Treat. 2015 Dec;59:20-9. doi: 10.1016/j.jsat.2015.06.016. Epub 2015 Jul 3. PMID 26362000
- [Background] Barrington-Trimis JL, Braymiller JL, Unger JB, McConnell R, Stokes A, Leventhal AM, Sargent JD, Samet JM, Goodwin RD. Trends in the Age of Cigarette Smoking Initiation Among Young Adults in the US From 2002 to 2018. JAMA Netw Open. 2020 Oct 1;3(10):e2019022. doi: 10.1001/jamanetworkopen.2020.19022. PMID 33021650
- See also: Centers for Disease Control and Prevention. (2022). National Health Interview Survey. Centers for Disease Control and Prevention. — https://www.cdc.gov/nchs/nhis/index.html
- See also: National Academies of Sciences, Engineering, and Medicine. (2018). Public health consequences of e-cigarettes. The National Academies Press. — https://nap.nationalacademies.org/catalog/24952/public-health-consequences-of-e-cigarettes
- See also: National Center for Chronic Disease Prevention and Health Promotion (US) Office on Smoking and Health. (2014). Patterns of tobacco use among U.S. youth, young adults, and adults. The Health Consequences of Smoking-50 Years of Progress: A Report of the Su — https://www.ncbi.nlm.nih.gov/books/NBK294302/
- See also: National Substance Use and Mental Health Services Survey (N-SUMHSS) release (2022). SAMHSA.gov. (2022). — https://www.samhsa.gov/data/data-we-collect/n-sumhss-national-substance-use-and-mental-health-services-survey/annual-releases/2022
- See also: Substance Abuse and Mental Health Services Administration. (2023). Mental Health for Young Adults. — https://www.samhsa.gov/mental-health/children-and-families/young-adults
- See also: U.S. Department of Health and Human Services. (2023). Do people with mental illness and substance use disorders use tobacco more often?. National Institutes of Health. — https://nida.nih.gov/publications/research-reports/tobacco-nicotine-e-cigarettes/do-people-mental-illness-substance-use-disorders-use-tobacco-more-often
- See also: U.S. initiatives. Campaign for Tobacco-Free Kids. (2025). — https://www.tobaccofreekids.org/what-we-do/us
- See also: World Health Organization. (2023 a). Tobacco fact sheet. World Health Organization. — https://www.who.int/news-room/fact-sheets/detail/tobacco